CLINICAL TRIAL: NCT01054820
Title: Multicenter, Open-Label Study to Assess the Effectiveness and Safety of FLECTOR Patch for Treatment of Acute Back Strain
Brief Title: Study to Assess the Effectiveness and Safety of FLECTOR Patch for Treatment of Acute Back Strain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K353-09-4001; B4811001
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-07

CONDITIONS: Acute Back Strain
Keywords: FLECTORÂ® Patch; acute back strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLECTORA Patch (diclofenac epolamine topical patch) 1.3% (Experimental): One patch applied every 12 hours
  Interventions: Drug: FLECTORÂ® Patch (diclofenac epolamine topical patch) 1.3%

INTERVENTIONS:
Drug: FLECTORÂ® Patch (diclofenac epolamine topical patch) 1.3% — One FLECTOR Patch applied to the most painful area on the subject's back every 12 hours for up to 14 days.

SUMMARY:
Although approved for minor strains, sprains and contusions, FLECTOR Patch has not been studied extensively in the setting of acute back strain. This study is being conducted as an initial step in demonstrating the benefit of FLECTOR Patch specifically for back strain. In particular, this study is expected to provide information about the amount of improvement in back strain among subjects using the FLECTOR Patch, which may then be used to inform subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

Participants in the study must:

1. have acute, non-radicular back strain with onset up to 10 days before the first visit
2. have intact, non-damaged skin at the proposed patch application site
3. be untreated or unresponsive to conservative pain treatment regimens and/or opioids
4. have a minimum pain intensity score of four (4) or more on a scale of 1-10 (a rating of zero (0) being "no pain" and a rating of ten (10) being "pain as bad as you can imagine")
5. have a normal neurologic examination

Exclusion Criteria:

Participants may not be in the study if they:

1. have had surgery or other chronic pain condition within 3 months before first treatment
2. have back pain radiating below the knee at time of enrollment
3. have neuropathic pain or have been treated with gabapentin or pregabalin for neuropathy
4. are being treated for or are known to currently have kidney or liver disease
5. have certain other diseases or are using certain types of other drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=K353-09-4001&StudyName=Study%20to%20Assess%20the%20Effectiveness%20and%20Safety%20of%20FLECTOR%20Patch%20for%20Treatment%20of%20Acute%20Back%20Strain

RESULTS

PARTICIPANT FLOW:
Groups:
- FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.: One patch applied topically every 12 hours for up to 14 days. Patch was to be applied at approximately the same time every day upon arising in the morning and at bedtime. The patch was to be applied to the most painful area to cover as much of the painful region as possible.
Period: Overall Study
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Started | 123
Completed | 121
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to End of Treatment (EOT) in Response to Modified Brief Pain Inventory (mBPI) Question 5: Average Pain Over the Last 24 Hours
Description: Participant-rated instrument to assess functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Question 5: Please rate your pain by marking the box beside the number that best describes your pain on the average (over the last 24 hours); rated on an 11 point Likert rating scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: Intent to Treat (ITT) population: had at least one application of FLECTOR® Patch, pain survey data at Baseline, and at least 1 follow-up visit. EOT score calculated by taking average of any non-missing scores recorded last 3 days of treatment; if no score on those days, EOT was single, most recent non-missing score recorded on a treatment day.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
scores on a scale
  Baseline | 6.46 (1.30)
  Change from baseline to EOT | -3.95 (2.51)
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Null hypothesis: no change from baseline. Study powered at 95 percent (%) to detect a mean change of at least 1.2 units, with assumed standard deviation of at most 3.2 units; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

2. Secondary Outcome: Number of Participants With Change From Baseline (Bsl) to EOT in Response to Modified Brief Pain Inventory (mBPI) Question 1: Pain Other Than Everyday Kind of Pain
Description: Participant-rated instrument to assess functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Question 1: Have you had pain other than everyday kinds of pain?; response = Yes or No.
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: ITT population; EOT score was the last non-missing score obtained on a treatment day, including the final treatment visit.
Measure: Number; unit: participants
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
participants
  Change at EOT: Bsl=Yes, EOT=Yes | 93
  Change at EOT: Bsl=Yes, EOT=No | 21
  Change at EOT: Bsl=No, EOT=Yes | 0
  Change at EOT: Bsl=No, EOT=No | 9
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Test type: Superiority or Other; p < 0.0001, McNemar — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

3. Secondary Outcome: Mean Change From Baseline to EOT in Response to Modified Brief Pain Inventory (mBPI) Question 3: Pain at Its Worst in the Last 24 Hours
Description: Participant-rated instrument to assess functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Question 3: Rate your pain at its worst in the last 24 hours; rated on an 11 point Likert rating scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: ITT population; EOT score calculated by taking average of any non-missing scores recorded last 3 days of treatment; if no score on those days, EOT was single, most recent non-missing score recorded on a treatment day.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
scores on a scale
  Baseline | 7.59 (1.19)
  Change from baseline to EOT | -4.50 (2.48)
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

4. Secondary Outcome: Mean Change From Baseline to EOT in Response to Modified Brief Pain Inventory (mBPI) Question 4: Pain at Its Least in the Last 24 Hours
Description: Participant-rated instrument to assess functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Question 4: Rate your pain at its least in the last 24 hours; rated on an 11 point Likert rating scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
scores on a scale
  Baseline | 5.46 (1.84)
  Change from baseline to EOT | -3.50 (2.30)
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

5. Secondary Outcome: Mean Change From Baseline to EOT in Response to Modified Brief Pain Inventory (mBPI) Question 6: Pain Right Now
Description: Participant-rated instrument to assess functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Question 6: Rate your pain right now; rated on an 11 point Likert rating scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
scores on a scale
  Baseline | 6.49 (1.76)
  Change from baseline to EOT | -4.28 (2.28)
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

6. Secondary Outcome: Mean Change From Baseline to EOT in Response to Modified Brief Pain Inventory (mBPI) Question 8: Percent Reduction in Pain From Baseline
Description: Participant-rated instrument to assess functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Question 8: Rate your percent reduction in pain from Baseline (0% = no relief to 100% = complete relief).
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: ITT population; EOT score calculated by taking average of any non-missing scores recorded last 3 days of treatment; if no score on those days, EOT was single, most recent non-missing score recorded on a treatment day. N=number of participants with analyzable data for Question 8 at observation.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 119
percent
  Baseline | 2.94 (11.23)
  Change from baseline to EOT | 67.30 (30.58)
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

7. Secondary Outcome: Number of Participants Per Global Pain Relief Scores at the End of Treatment as Assessed by the Participant
Description: Global pain relief as assessed by participant using a 5-point scale where 5 = complete relief, 4=a lot of improvement, 3=moderate improvement, 2=slight improvement, and 1=no change.
Time Frame: End of Treatment (up to Day 15)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
participants
  5=Complete Relief | 53
  4=A Lot Of Improvement | 42
  3=Moderate Improvement | 12
  2=Slight Improvement | 12
  1=No Change | 4

8. Secondary Outcome: Number of Participants Per Global Pain Relief Scores at the End of Treatment as Assessed by the Investigator
Description: Participants' global pain relief as assessed by investigator using a 5-point scale where 5 = complete relief, 4=a lot of improvement, 3=moderate improvement, 2=slight improvement, and 1=no change.
Time Frame: End of Treatment (up to Day 15)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
participants
  5=Complete Relief | 58
  4=A Lot Of Improvement | 42
  3=Moderate Improvement | 8
  2=Slight Improvement | 10
  1=No Change | 5

9. Secondary Outcome: Mean Change From Baseline to EOT in Beck Depression Inventory® Il
Description: The Beck Depression Inventory® II consisted of 21 items, each with 4 categorical responses ranging from 0 (I do not feel sad) to 3 (I am so sad or unhappy that I can't stand it) with maximum possible score of 63; increase in the number reflected an increase in severity. Total Beck Depression Inventory® II scores classified as follows: 1 to 10=normal ups and downs; 11 to 16=mild mood disturbance; 17 to 20=borderline clinical depression; 21 to 30=moderate depression; 31 to 40=severe depression; and >40=extreme depression.
Time Frame: Baseline, End of Treatment (last visit up to Day 15)
Population: ITT population; End-of-Treatment score was the most recent non-missing value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
scores on a scale
  Baseline | 3.44 (5.47)
  Change from baseline to EOT | -1.54 (3.05)
Statistical Analysis 1: Comparison: FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05

10. Secondary Outcome: Number of Participants Per Patch Satisfaction Response at the End of Treatment as Assessed by Participant
Description: Participant satisfaction with the FLECTOR® Patch rated on a 5-point scale scored as 5=Very Satisfied, 4=Satisfied, 3=No Preference, 2=Dissatisfied, and 1=Very Dissatisfied.
Time Frame: End of Treatment (last visit up to Day 15)
Population: ITT; End-of-Treatment score for patch satisfaction consisted of the last value recorded.
Measure: Number; unit: participants
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
participants
  5=Very Satisfied | 63
  4=Satisfied | 45
  3=No Preference | 6
  2=Dissatisfied | 8
  1=Very Dissatisfied | 1

11. Secondary Outcome: Number of Participants Per Patch Satisfaction Response at the End of Treatment as Assessed by the Investigator
Description: Investigator's assessment of participants' satisfaction with the FLECTOR® Patch rated on a 5-point scale scored as 5=Very Satisfied, 4=Satisfied, 3=No Preference, 2=Dissatisfied, and 1=Very Dissatisfied.
Time Frame: End of Treatment (last visit up to Day 15)
Population: ITT; End-of-Treatment score for patch satisfaction consisted of the last value recorded.
Measure: Number; unit: participants
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Number analyzed (Participants) | 123
participants
  5=Very Satisfied | 66
  4=Satisfied | 39
  3=No Preference | 9
  2=Dissatisfied | 8
  1=Very Dissatisfied | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 14 days after last dose. Adverse events ongoing at the last visit were to be followed until resolution or until no further follow-up warranted.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%.
Serious Adverse Events (participants affected / at risk) | 1/123
Other Adverse Events (participants affected / at risk) | 15/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%. (N=123)
Non-cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLECTOR® Patch (Diclofenac Epolamine Topical Patch) 1.3%. (N=123)
Tachycardia (Cardiac disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Application site rash (Injury, poisoning and procedural complications) | 3
Application site pruritus (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.